CLINICAL TRIAL: NCT07015567
Title: Contextualised, Culture-sensitive Diagnosis and Psychotherapy for the Treatment of Complex Post-traumatic Stress Disorder Among Displaced People in Switzerland and Germany: A Two-step Multicentric Randomised Clinical Trial
Brief Title: Treatment of Complex Post-traumatic Stress Disorder Among Displaced People in Switzerland and Germany
Acronym: ESTAIR_REFUGEE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eva Heim (Other)
Responsible Party: Sponsor-Investigator, Eva Heim, Associate professor, University of Lausanne
Organization: University of Lausanne (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: BASEC 2025-00450; 10001G_212438 (Other Grant/Funding Number: Swiss National Science Foundation)
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Complex Post-Traumatic Stress Disorder
Keywords: Refugee populations; Cultural adaptation; Factorial experiment; Culturally sensitive psychotherapy

STUDY DESIGN:
Intervention Model Description: In this single-blind randomised trial, the study team will use a Balanced Incomplete Block Design (BIBD), which corresponds to an incomplete factorial experiment. The design encompasses 48 experimental conditions, where all participants will receive three out of four modules of the adapted ESTAIR manual and will have one waiting period (at the start or at the end of their treatment). The investigators will test all possible combinations and sequences of these modules. Assessments (between modules and after the last module) will be conducted by assessors. Assessors will not have access to the experimental condition to which the participant is assigned, nor to any information related to the therapy process.
Who Masked: Outcomes Assessor
Masking Description: Independent assessors are blinded to the intervention compoments (i.e., module or waiting) participants have received.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (48):
- 1. Waiting period, emotion regulation, negative self-concept, interpersonal relationships (Experimental)
  Interventions: Behavioral: Emotion regulation module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Negative self-concept module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Interpersonal relationships module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET)
- 2. Waiting period, emotion regulation, negative self-concept, narrative exposure therapy (Experimental)
  Interventions: Behavioral: Emotion regulation module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Negative self-concept module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Narrative exposure therapy module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET)
- 3. Waiting period, emotion regulation, interpersonal relationships, negative self-concept (Experimental)
  Interventions: Behavioral: Emotion regulation module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Negative self-concept module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Interpersonal relationships module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET)
- 4. Waiting period, emotion regulation, interpersonal relationships, narrative exposure therapy (Experimental)
  Interventions: Behavioral: Emotion regulation module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Interpersonal relationships module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Narrative exposure therapy module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET)
- 5. Waiting period, emotion regulation, narrative exposure therapy, negative self-concept (Experimental)
  Interventions: Behavioral: Emotion regulation module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Negative self-concept module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Narrative exposure therapy module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET)
- 6. Waiting period, emotion regulation, narrative exposure therapy, interpersonal relationships (Experimental)
  Interventions: Behavioral: Emotion regulation module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Interpersonal relationships module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Narrative exposure therapy module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET)
- 7. Waiting period, negative self-concept, emotion regulation, interpersonal relationships (Experimental)
  Interventions: Behavioral: Emotion regulation module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Negative self-concept module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Interpersonal relationships module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET)
- 8. Waiting period, negative self-concept, emotion regulation, narrative exposure therapy (Experimental)
  Interventions: Behavioral: Emotion regulation module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Negative self-concept module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Narrative exposure therapy module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET)
- 9. Waiting period, negative self-concept, interpersonal relationships, emotion regulation (Experimental)
  Interventions: Behavioral: Emotion regulation module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Negative self-concept module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Interpersonal relationships module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET)
- 10. Waiting period, negative self-concept, interpersonal relationships, narrative exposure therapy (Experimental)
  Interventions: Behavioral: Negative self-concept module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Interpersonal relationships module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Narrative exposure therapy module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET)
- 11. Waiting period, negative self-concept, narrative exposure therapy, emotion regulation (Experimental)
  Interventions: Behavioral: Emotion regulation module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Negative self-concept module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Narrative exposure therapy module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET)
- 12. Waiting period, negative self-concept, narrative exposure therapy, interpersonal relationships (Experimental)
  Interventions: Behavioral: Negative self-concept module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Interpersonal relationships module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Narrative exposure therapy module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET)
- 13. Waiting period, interpersonal relationships, emotion regulation, negative self-concept (Experimental)
  Interventions: Behavioral: Emotion regulation module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Negative self-concept module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Interpersonal relationships module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET)
- 14. Waiting period, interpersonal relationships, emotion regulation, narrative exposure therapy (Experimental)
  Interventions: Behavioral: Emotion regulation module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Interpersonal relationships module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Narrative exposure therapy module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET)
- 15. Waiting period, interpersonal relationships, negative self-concept, emotion regulation (Experimental)
  Interventions: Behavioral: Emotion regulation module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Negative self-concept module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Interpersonal relationships module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET)
- 16. Waiting period, interpersonal relationships, negative self-concept, narrative exposure therapy (Experimental)
  Interventions: Behavioral: Negative self-concept module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Interpersonal relationships module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Narrative exposure therapy module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET)
- 17. Waiting period, interpersonal relationships, narrative exposure therapy, emotion regulation (Experimental)
  Interventions: Behavioral: Emotion regulation module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Interpersonal relationships module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Narrative exposure therapy module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET)
- 18. Waiting period, interpersonal relationships, narrative exposure therapy, negative self-concept (Experimental)
  Interventions: Behavioral: Negative self-concept module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Interpersonal relationships module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Narrative exposure therapy module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET)
- 19. Waiting period, narrative exposure therapy, emotion regulation, negative self-concept (Experimental)
  Interventions: Behavioral: Emotion regulation module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Negative self-concept module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Narrative exposure therapy module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET)
- 20. Waiting period, narrative exposure therapy, emotion regulation, interpersonal relationships (Experimental)
  Interventions: Behavioral: Emotion regulation module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Interpersonal relationships module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Narrative exposure therapy module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET)
- 21. Waiting period, narrative exposure therapy, negative self-concept, emotion regulation (Experimental)
  Interventions: Behavioral: Emotion regulation module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Negative self-concept module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Narrative exposure therapy module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET)
- 22. Waiting period, narrative exposure therapy, negative self-concept, interpersonal relationships (Experimental)
  Interventions: Behavioral: Negative self-concept module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Interpersonal relationships module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Narrative exposure therapy module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET)
- 23. Waiting period, narrative exposure therapy, interpersonal relationships, emotion regulation (Experimental)
  Interventions: Behavioral: Emotion regulation module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Interpersonal relationships module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Narrative exposure therapy module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET)
- 24. Waiting period, narrative exposure therapy, interpersonal relationships, negative self-concept (Experimental)
  Interventions: Behavioral: Negative self-concept module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Interpersonal relationships module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Narrative exposure therapy module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET)
- 25. Emotion regulation, negative self-concept, interpersonal relationships, waiting period (Experimental)
  Interventions: Behavioral: Emotion regulation module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Negative self-concept module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Interpersonal relationships module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET)
- 26. Emotion regulation, negative self-concept, narrative exposure therapy, waiting period (Experimental)
  Interventions: Behavioral: Emotion regulation module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Negative self-concept module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Narrative exposure therapy module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET)
- 27. Emotion regulation, interpersonal relationships, negative self-concept, waiting period (Experimental)
  Interventions: Behavioral: Emotion regulation module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Negative self-concept module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Interpersonal relationships module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET)
- 28. Emotion regulation, interpersonal relationships, narrative exposure therapy, waiting period (Experimental)
  Interventions: Behavioral: Emotion regulation module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Interpersonal relationships module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Narrative exposure therapy module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET)
- 29. Emotion regulation, narrative exposure therapy, negative self-concept, waiting period (Experimental)
  Interventions: Behavioral: Emotion regulation module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Negative self-concept module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Narrative exposure therapy module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET)
- 30. Emotion regulation, narrative exposure therapy, interpersonal relationships, waiting period (Experimental)
  Interventions: Behavioral: Emotion regulation module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Interpersonal relationships module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Narrative exposure therapy module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET)
- 31. Negative self-concept, emotion regulation, interpersonal relationships, waiting period (Experimental)
  Interventions: Behavioral: Emotion regulation module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Negative self-concept module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Interpersonal relationships module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET)
- 32. Negative self-concept, emotion regulation, narrative exposure therapy, waiting period (Experimental)
  Interventions: Behavioral: Emotion regulation module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Negative self-concept module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Narrative exposure therapy module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET)
- 33. Negative self-concept, interpersonal relationships, emotion regulation, waiting period (Experimental)
  Interventions: Behavioral: Emotion regulation module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Negative self-concept module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Interpersonal relationships module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET)
- 34. Negative self-concept, interpersonal relationships, narrative exposure therapy, waiting period (Experimental)
  Interventions: Behavioral: Negative self-concept module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Interpersonal relationships module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Narrative exposure therapy module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET)
- 35. Negative self-concept, narrative exposure therapy, emotion regulation, waiting period (Experimental)
  Interventions: Behavioral: Emotion regulation module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Negative self-concept module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Narrative exposure therapy module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET)
- 36. Negative self-concept, narrative exposure therapy, interpersonal relationships, waiting period (Experimental)
  Interventions: Behavioral: Negative self-concept module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Interpersonal relationships module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Narrative exposure therapy module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET)
- 37. Interpersonal relationships, emotion regulation, negative self-concept, waiting period (Experimental)
  Interventions: Behavioral: Emotion regulation module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Negative self-concept module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Interpersonal relationships module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET)
- 38. Interpersonal relationships, emotion regulation, narrative exposure therapy, waiting period (Experimental)
  Interventions: Behavioral: Emotion regulation module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Interpersonal relationships module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Narrative exposure therapy module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET)
- 39. Interpersonal relationships, negative self-concept, emotion regulation, waiting period (Experimental)
  Interventions: Behavioral: Emotion regulation module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Negative self-concept module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Interpersonal relationships module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET)
- 40. Interpersonal relationships, negative self-concept, narrative exposure therapy, waiting period (Experimental)
  Interventions: Behavioral: Negative self-concept module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Interpersonal relationships module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Narrative exposure therapy module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET)
- 41. Interpersonal relationships, narrative exposure therapy, emotion regulation, waiting period (Experimental)
  Interventions: Behavioral: Emotion regulation module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Interpersonal relationships module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Narrative exposure therapy module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET)
- 42. Interpersonal relationships, narrative exposure therapy, negative self-concept, waiting period (Experimental)
  Interventions: Behavioral: Negative self-concept module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Interpersonal relationships module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Narrative exposure therapy module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET)
- 43. Narrative exposure therapy, emotion regulation, negative self-concept, waiting period (Experimental)
  Interventions: Behavioral: Emotion regulation module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Negative self-concept module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Narrative exposure therapy module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET)
- 44. Narrative exposure therapy, emotion regulation, interpersonal relationships, waiting period (Experimental)
  Interventions: Behavioral: Emotion regulation module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Interpersonal relationships module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Narrative exposure therapy module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET)
- 45. Narrative exposure therapy, negative self-concept, emotion regulation, waiting period (Experimental)
  Interventions: Behavioral: Emotion regulation module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Negative self-concept module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Narrative exposure therapy module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET)
- 46. Narrative exposure therapy, negative self-concept, interpersonal relationships, waiting period (Experimental)
  Interventions: Behavioral: Negative self-concept module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Interpersonal relationships module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Narrative exposure therapy module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET)
- 47. Narrative exposure therapy, interpersonal relationships, emotion regulation, waiting period (Experimental)
  Interventions: Behavioral: Emotion regulation module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Interpersonal relationships module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Narrative exposure therapy module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET)
- 48. Narrative exposure therapy, interpersonal relationships, negative self-concept, waiting period (Experimental)
  Interventions: Behavioral: Negative self-concept module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Interpersonal relationships module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET); Behavioral: Narrative exposure therapy module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET)

INTERVENTIONS:
Behavioral: Emotion regulation module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET) — ESTAIR is a psychotherapeutic manual for the treatment of CPTSD. The manual was adapted to the target population. It contains 24 sessions which are organised in four modules, including a module about emotion regulation. This module contains exercises for emotional awareness and emotion regulation with different focuses (on body, thoughts and behaviour).
  Arms: 1. Waiting period, emotion regulation, negative self-concept, interpersonal relationships; 11. Waiting period, negative self-concept, narrative exposure therapy, emotion regulation; 13. Waiting period, interpersonal relationships, emotion regulation, negative self-concept; 14. Waiting period, interpersonal relationships, emotion regulation, narrative exposure therapy; 15. Waiting period, interpersonal relationships, negative self-concept, emotion regulation; 17. Waiting period, interpersonal relationships, narrative exposure therapy, emotion regulation; 19. Waiting period, narrative exposure therapy, emotion regulation, negative self-concept; 2. Waiting period, emotion regulation, negative self-concept, narrative exposure therapy; 20. Waiting period, narrative exposure therapy, emotion regulation, interpersonal relationships; 21. Waiting period, narrative exposure therapy, negative self-concept, emotion regulation; 23. Waiting period, narrative exposure therapy, interpersonal relationships, emotion regulation; 25. Emotion regulation, negative self-concept, interpersonal relationships, waiting period; 26. Emotion regulation, negative self-concept, narrative exposure therapy, waiting period; 27. Emotion regulation, interpersonal relationships, negative self-concept, waiting period; 28. Emotion regulation, interpersonal relationships, narrative exposure therapy, waiting period; 29. Emotion regulation, narrative exposure therapy, negative self-concept, waiting period; 3. Waiting period, emotion regulation, interpersonal relationships, negative self-concept; 30. Emotion regulation, narrative exposure therapy, interpersonal relationships, waiting period; 31. Negative self-concept, emotion regulation, interpersonal relationships, waiting period; 32. Negative self-concept, emotion regulation, narrative exposure therapy, waiting period; 33. Negative self-concept, interpersonal relationships, emotion regulation, waiting period; 35. Negative self-concept, narrative exposure therapy, emotion regulation, waiting period; 37. Interpersonal relationships, emotion regulation, negative self-concept, waiting period; 38. Interpersonal relationships, emotion regulation, narrative exposure therapy, waiting period; 39. Interpersonal relationships, negative self-concept, emotion regulation, waiting period; 4. Waiting period, emotion regulation, interpersonal relationships, narrative exposure therapy; 41. Interpersonal relationships, narrative exposure therapy, emotion regulation, waiting period; 43. Narrative exposure therapy, emotion regulation, negative self-concept, waiting period; 44. Narrative exposure therapy, emotion regulation, interpersonal relationships, waiting period; 45. Narrative exposure therapy, negative self-concept, emotion regulation, waiting period; 47. Narrative exposure therapy, interpersonal relationships, emotion regulation, waiting period; 5. Waiting period, emotion regulation, narrative exposure therapy, negative self-concept; 6. Waiting period, emotion regulation, narrative exposure therapy, interpersonal relationships; 7. Waiting period, negative self-concept, emotion regulation, interpersonal relationships; 8. Waiting period, negative self-concept, emotion regulation, narrative exposure therapy; 9. Waiting period, negative self-concept, interpersonal relationships, emotion regulation
Behavioral: Negative self-concept module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET) — ESTAIR is a psychotherapeutic manual for the treatment of CPTSD. The manual was adapted to the target population. It contains 24 sessions which are organised in four modules, including a module about negative self-concept. In this module, the manual tackles topics such as what is the self, thinking about the self through cognitive restructuring, criticism and compassion and the self in relation to others.
  Arms: 1. Waiting period, emotion regulation, negative self-concept, interpersonal relationships; 10. Waiting period, negative self-concept, interpersonal relationships, narrative exposure therapy; 11. Waiting period, negative self-concept, narrative exposure therapy, emotion regulation; 12. Waiting period, negative self-concept, narrative exposure therapy, interpersonal relationships; 13. Waiting period, interpersonal relationships, emotion regulation, negative self-concept; 15. Waiting period, interpersonal relationships, negative self-concept, emotion regulation; 16. Waiting period, interpersonal relationships, negative self-concept, narrative exposure therapy; 18. Waiting period, interpersonal relationships, narrative exposure therapy, negative self-concept; 19. Waiting period, narrative exposure therapy, emotion regulation, negative self-concept; 2. Waiting period, emotion regulation, negative self-concept, narrative exposure therapy; 21. Waiting period, narrative exposure therapy, negative self-concept, emotion regulation; 22. Waiting period, narrative exposure therapy, negative self-concept, interpersonal relationships; 24. Waiting period, narrative exposure therapy, interpersonal relationships, negative self-concept; 25. Emotion regulation, negative self-concept, interpersonal relationships, waiting period; 26. Emotion regulation, negative self-concept, narrative exposure therapy, waiting period; 27. Emotion regulation, interpersonal relationships, negative self-concept, waiting period; 29. Emotion regulation, narrative exposure therapy, negative self-concept, waiting period; 3. Waiting period, emotion regulation, interpersonal relationships, negative self-concept; 31. Negative self-concept, emotion regulation, interpersonal relationships, waiting period; 32. Negative self-concept, emotion regulation, narrative exposure therapy, waiting period; 33. Negative self-concept, interpersonal relationships, emotion regulation, waiting period; 34. Negative self-concept, interpersonal relationships, narrative exposure therapy, waiting period; 35. Negative self-concept, narrative exposure therapy, emotion regulation, waiting period; 36. Negative self-concept, narrative exposure therapy, interpersonal relationships, waiting period; 37. Interpersonal relationships, emotion regulation, negative self-concept, waiting period; 39. Interpersonal relationships, negative self-concept, emotion regulation, waiting period; 40. Interpersonal relationships, negative self-concept, narrative exposure therapy, waiting period; 42. Interpersonal relationships, narrative exposure therapy, negative self-concept, waiting period; 43. Narrative exposure therapy, emotion regulation, negative self-concept, waiting period; 45. Narrative exposure therapy, negative self-concept, emotion regulation, waiting period; 46. Narrative exposure therapy, negative self-concept, interpersonal relationships, waiting period; 48. Narrative exposure therapy, interpersonal relationships, negative self-concept, waiting period; 5. Waiting period, emotion regulation, narrative exposure therapy, negative self-concept; 7. Waiting period, negative self-concept, emotion regulation, interpersonal relationships; 8. Waiting period, negative self-concept, emotion regulation, narrative exposure therapy; 9. Waiting period, negative self-concept, interpersonal relationships, emotion regulation
Behavioral: Interpersonal relationships module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET) — ESTAIR is a psychotherapeutic manual for the treatment of CPTSD. The manual was adapted to the target population. It contains 24 sessions which are organised in four modules, including a module about interpersonal relationships. This module includes exercises to understand relationship patterns, increasing assertiveness, practicing assertiveness, and managing power.
  Arms: 1. Waiting period, emotion regulation, negative self-concept, interpersonal relationships; 10. Waiting period, negative self-concept, interpersonal relationships, narrative exposure therapy; 12. Waiting period, negative self-concept, narrative exposure therapy, interpersonal relationships; 13. Waiting period, interpersonal relationships, emotion regulation, negative self-concept; 14. Waiting period, interpersonal relationships, emotion regulation, narrative exposure therapy; 15. Waiting period, interpersonal relationships, negative self-concept, emotion regulation; 16. Waiting period, interpersonal relationships, negative self-concept, narrative exposure therapy; 17. Waiting period, interpersonal relationships, narrative exposure therapy, emotion regulation; 18. Waiting period, interpersonal relationships, narrative exposure therapy, negative self-concept; 20. Waiting period, narrative exposure therapy, emotion regulation, interpersonal relationships; 22. Waiting period, narrative exposure therapy, negative self-concept, interpersonal relationships; 23. Waiting period, narrative exposure therapy, interpersonal relationships, emotion regulation; 24. Waiting period, narrative exposure therapy, interpersonal relationships, negative self-concept; 25. Emotion regulation, negative self-concept, interpersonal relationships, waiting period; 27. Emotion regulation, interpersonal relationships, negative self-concept, waiting period; 28. Emotion regulation, interpersonal relationships, narrative exposure therapy, waiting period; 3. Waiting period, emotion regulation, interpersonal relationships, negative self-concept; 30. Emotion regulation, narrative exposure therapy, interpersonal relationships, waiting period; 31. Negative self-concept, emotion regulation, interpersonal relationships, waiting period; 33. Negative self-concept, interpersonal relationships, emotion regulation, waiting period; 34. Negative self-concept, interpersonal relationships, narrative exposure therapy, waiting period; 36. Negative self-concept, narrative exposure therapy, interpersonal relationships, waiting period; 37. Interpersonal relationships, emotion regulation, negative self-concept, waiting period; 38. Interpersonal relationships, emotion regulation, narrative exposure therapy, waiting period; 39. Interpersonal relationships, negative self-concept, emotion regulation, waiting period; 4. Waiting period, emotion regulation, interpersonal relationships, narrative exposure therapy; 40. Interpersonal relationships, negative self-concept, narrative exposure therapy, waiting period; 41. Interpersonal relationships, narrative exposure therapy, emotion regulation, waiting period; 42. Interpersonal relationships, narrative exposure therapy, negative self-concept, waiting period; 44. Narrative exposure therapy, emotion regulation, interpersonal relationships, waiting period; 46. Narrative exposure therapy, negative self-concept, interpersonal relationships, waiting period; 47. Narrative exposure therapy, interpersonal relationships, emotion regulation, waiting period; 48. Narrative exposure therapy, interpersonal relationships, negative self-concept, waiting period; 6. Waiting period, emotion regulation, narrative exposure therapy, interpersonal relationships; 7. Waiting period, negative self-concept, emotion regulation, interpersonal relationships; 9. Waiting period, negative self-concept, interpersonal relationships, emotion regulation
Behavioral: Narrative exposure therapy module of Enhanced Skills Training in Affective and Interpersonal Regulation combined with Narrative Exposure Therapy (ESTAIR/NET) — ESTAIR is a psychotherapeutic manual for the treatment of CPTSD. It contains 24 sessions which are organised in four modules. The manual was adapted to the target population. In this context, the module "modified prolonged exposure" was replaced with Narrative Exposure Therapy (NET). NET is a standardised approach for the treatment of PTSD that has been tested across diverse social and cultural contexts. In this intervention, patients and therapists elaborate together a chronological timeline (called "the lifeline") of patient's life and the traumatic events, using a rope, stones for traumatic events, and flowers for positive events. Thereafter, the traumatic events are discussed in detail, one in each session. At the end of each session, patients receive a written form of these narrations, co-signed by patient and the therapist.
  Arms: 10. Waiting period, negative self-concept, interpersonal relationships, narrative exposure therapy; 11. Waiting period, negative self-concept, narrative exposure therapy, emotion regulation; 12. Waiting period, negative self-concept, narrative exposure therapy, interpersonal relationships; 14. Waiting period, interpersonal relationships, emotion regulation, narrative exposure therapy; 16. Waiting period, interpersonal relationships, negative self-concept, narrative exposure therapy; 17. Waiting period, interpersonal relationships, narrative exposure therapy, emotion regulation; 18. Waiting period, interpersonal relationships, narrative exposure therapy, negative self-concept; 19. Waiting period, narrative exposure therapy, emotion regulation, negative self-concept; 2. Waiting period, emotion regulation, negative self-concept, narrative exposure therapy; 20. Waiting period, narrative exposure therapy, emotion regulation, interpersonal relationships; 21. Waiting period, narrative exposure therapy, negative self-concept, emotion regulation; 22. Waiting period, narrative exposure therapy, negative self-concept, interpersonal relationships; 23. Waiting period, narrative exposure therapy, interpersonal relationships, emotion regulation; 24. Waiting period, narrative exposure therapy, interpersonal relationships, negative self-concept; 26. Emotion regulation, negative self-concept, narrative exposure therapy, waiting period; 28. Emotion regulation, interpersonal relationships, narrative exposure therapy, waiting period; 29. Emotion regulation, narrative exposure therapy, negative self-concept, waiting period; 30. Emotion regulation, narrative exposure therapy, interpersonal relationships, waiting period; 32. Negative self-concept, emotion regulation, narrative exposure therapy, waiting period; 34. Negative self-concept, interpersonal relationships, narrative exposure therapy, waiting period; 35. Negative self-concept, narrative exposure therapy, emotion regulation, waiting period; 36. Negative self-concept, narrative exposure therapy, interpersonal relationships, waiting period; 38. Interpersonal relationships, emotion regulation, narrative exposure therapy, waiting period; 4. Waiting period, emotion regulation, interpersonal relationships, narrative exposure therapy; 40. Interpersonal relationships, negative self-concept, narrative exposure therapy, waiting period; 41. Interpersonal relationships, narrative exposure therapy, emotion regulation, waiting period; 42. Interpersonal relationships, narrative exposure therapy, negative self-concept, waiting period; 43. Narrative exposure therapy, emotion regulation, negative self-concept, waiting period; 44. Narrative exposure therapy, emotion regulation, interpersonal relationships, waiting period; 45. Narrative exposure therapy, negative self-concept, emotion regulation, waiting period; 46. Narrative exposure therapy, negative self-concept, interpersonal relationships, waiting period; 47. Narrative exposure therapy, interpersonal relationships, emotion regulation, waiting period; 48. Narrative exposure therapy, interpersonal relationships, negative self-concept, waiting period; 5. Waiting period, emotion regulation, narrative exposure therapy, negative self-concept; 6. Waiting period, emotion regulation, narrative exposure therapy, interpersonal relationships; 8. Waiting period, negative self-concept, emotion regulation, narrative exposure therapy

SUMMARY:
In WHO ICD-11 (its latest edition), the diagnostic criteria for post-traumatic stress disorder (PTSD) were revised, and a new sibling disorder, complex post-traumatic stress disorder (CPTSD) was introduced. CPTSD is a debilitating condition associated with severe, prolonged, or chronic trauma. Refugee populations are affected by high prevalence of CPTSD because of high rates of such trauma (e.g. torture). Untreated CPTSD has negative consequences for quality of life and for integration into the host society. Evidence indicates cultural variation in the phenomenology of CPTSD.

Modular approaches, e.g., the Skills Training in Affective and Interpersonal Regulation combined with Modified Prolonged Exposure (ESTAIR/MPE), have been recommended for the treatment of CPTSD. However, they have not been tested in a clinical trial among refugees so far and there are no available publications about their effectiveness in CPTSD symptom reduction among this population. Research suggests a higher symptom reduction of trauma-focused techniques, such as Narrative Exposure Therapy (NET), among refugee population. In a previous study, the investigators pilot tested a version of ESTAIR/NET that was adapted to sociocultural and structural aspects related to psychopathology in refugee populations. The performance of these culturally adapted modules in CPTSD symptom reduction among the refugee population remains to be assessed.

The present clinical trial seeks to assess the effect of the culturally adapted modules of the ESTAIR manual on symptom reduction among refugees and asylum seekers diagnosed with CPTSD.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signature
* Refugees and asylum seekers with a valid residence permit (N, F, B, or C status)
* Speaking Arabic, Farsi/Dari, Pashtu, Kurdish (different dialects), or Turkish
* A psychotherapy is indicated and was prescribed
* Participated to part 1 of the study and was diagnosed with CPTSD on the basis of the standard International Trauma Interview and the Socio-cultural and structural addendum (SCSA). The diagnosis is done based on the clinical judgement by the local therapist.

Exclusion Criteria:

* Acute psychosis
* Imminent risk of suicide
* Severe alcohol and/or substance abuse
* Being enrolled in another psychotherapy
* Inability to follow study procedures (i.e., cognitive impairment)
* Inability to give informed consent
* Known pregnancy

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2026-01-21 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
CPTSD symptom change | 8 months
  CPTSD symptom change will be assessed with the International Trauma Questionnaire (ITQ-28). This questionnaire contains 28 items on symptoms that are self-rated on a Likert scale of 0-4, with a maximum total score of 112.

SECONDARY OUTCOMES:
Depression | 8 months
  Patient Health Questionnaire (PHQ-9). The PHQ-9 score may range from 0 to 27, since each of the 9 items can be scored from 0 (not at all) to 3 (nearly every day). Higher scores mean higher levels of depression.
Anxiety | 8 months
  General Anxiety Disorder Questionnaire (GAD-7). The GAD-7 score may range from 0 to 21, since each of the 7 items can be scored from 0 (not at all) to 3 (nearly every day). Higher scores mean higher levels of anxiety.
Somatic symptoms | 8 months
  Somatic Symptoms Scale (SSS-8). The SSS-8 score may range from 0 to 32, since each of the 8 items can be scored from 0 (not at all) to 4 (severely). Higher scores mean higher levels of somatic symptoms.
Well-being | 8 months
  WHO-5 questionnaire. Scores range from 0-25, with higher scores reflecting higher levels of well-being.
Dissociative symptoms (Shut-D) | 8 months
  The Shut-D contains 13 items measuring dissociative symptoms such as fainting or analgesia. Each item is rated on a scale from 0 to 3. The total score ranges from 0 to 39.

CONTACTS AND LOCATIONS:
Locations (7):
- Centra, Hamburg, Hamburg, Germany
- Switzerland (6):
  - Psychiatrie Basel-Land, Liestal, Basel-Landschaft
  - Psy4Asyl, Aarau, Canton of Aargau
  - UPK Transkulturelle Ambulanz, Basel, Canton of Basel-City
  - SRK Ambulatorium für Folter- und Kriegsopfer, Wabern, Canton of Bern
  - Appartenances - CPM Lausanne, Lausanne, Canton of Vaud
  - Appartenances - CPM Yverdon-les-Bains, Yverdon-les-Bains, Canton of Vaud

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Heim E, Karatzias T, Maercker A. Cultural concepts of distress and complex PTSD: Future directions for research and treatment. Clin Psychol Rev. 2022 Apr;93:102143. doi: 10.1016/j.cpr.2022.102143. Epub 2022 Mar 7. PMID 35313215
- See also: HumRes is the Federal Office of Public Health's website for the general public on human research in Switzerland — https://www.humanforschung-schweiz.ch/de/